CLINICAL TRIAL: NCT00442013
Title: Phase III: The Study of Acid Reflux in Children With Asthma
Brief Title: Lansoprazole to Treat Children With Asthma
Acronym: SARCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Lung Association Asthma Clinical Research Centers (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Janet Holbrook, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 454; U01HL080450-01 (NIH); NCT00604851 (obsolete NCT alias)
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Results first posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lansoprazole (Experimental): Participants in this group will receive lansoprazole on a daily basis for 6 months. There are two doses of Lansoprazole solutab provided to participants depending on participant body weight at randomization: 1.) less than 30kg will receive 15mg po once daily or 2.)greater or equal to 30kg 30mg po once daily.
  Interventions: Drug: Lansoprazole
- Matching placebo (Placebo Comparator): Participants in this group will receive a matching placebo on a daily basis for 6 months. To maintain masking, there are two doses of the matching placebo provided to participants depending on participant body weight at randomization: 1.) less than 30kg will receive 15mg po once daily or 2.)greater or equal to 30kg 30mg po once daily.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Lansoprazole — Participants less than 30 kg will receive 15 mg a day, by mouth; participants greater than or equal to 30 kg will receive 30 mg a day, by mouth.
  Other Names: Prevacid
  Arms: Lansoprazole
Drug: Matching placebo — Participants will receive a placebo pill on a daily basis. To maintain masking, there are two doses of the matching placebo provided to participants depending on participant body weight at randomization: 1.) less than 30kg will receive 15mg po once daily or 2.)greater or equal to 30kg 30mg po once daily.
  Other Names: Matching placebo manufactured by TAP Pharmaceuticals
  Arms: Matching placebo

SUMMARY:
Many individuals with asthma also experience gastroesophageal reflux disease (GERD), a condition in which excess stomach acid flows backwards into the esophagus. This study will evaluate the effectiveness of lansoprazole, a medication commonly used to treat GERD in improving asthma control and reducing symptoms in children with poorly controlled asthma.

DETAILED DESCRIPTION:
Approximately 75% of individuals with asthma also experience GERD. If left untreated, GERD can lead to lung damage, esophageal ulcers, or esophageal cancer. Children and adults whose asthma is poorly controlled with inhaled corticosteroids are often prescribed drugs that suppress gastric acid production; however, this treatment is expensive and has not been proven beneficial. Lansoprazole is a proton pump inhibitor medication that reduces stomach acid production. It may also decrease the frequency of asthma exacerbations in children with poorly controlled asthma. The purpose of this study is to evaluate the effectiveness of lansoprazole at improving asthma control, quality of life, and lung function in children with asthma.

This study will enroll children with poor asthma control who are receiving inhaled corticosteroids. Participants will be randomly assigned to receive either lansoprazole or placebo on a daily basis for 6 months. Study visits will occur at baseline and Weeks 4, 8, 12, 16, 20, and 24, and participants will be contacted by telephone at Week 2. A physical examination, blood collection, and methacholine challenge test will occur at selected visits. The methacholine challenge test will be used to help determine the severity of an individual's asthma. Lung function and airway pressure testing, questionnaires on asthma control and quality of life, medical history review, pill counts, and distribution of medication will occur at most study visits. Participants will record asthma symptoms and lung function in a daily diary throughout the study. A select group of participants will also wear an esophageal potential Hydrogen (pH) monitor for 24 hours to evaluate GERD symptoms and the relationship between GERD and asthma symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma
* At least one of the following lung function criteria must be documented in the year prior to study entry:

  1. Bronchial hyperresponsiveness confirmed by 12% or greater improvement in amount of air expired in first second during a forced expiratory maneuver (FEV1) post-bronchodilator, or
  2. Methacholine post-diluent baseline (PC20) less than 16 mg/ml, or
  3. Exercise bronchoprovocation test with at least a 20% decrease in FEV1
* Currently on stable dose of daily inhaled corticosteroid for asthma control (i.e., inhaled corticosteroid equivalent to 2 puffs of 44 ug twice per day [176 ug] of fluticasone or greater for 8 weeks or longer prior to study entry)
* Poor asthma control as defined by any one of the following criteria:

  1. Use of beta-agonist for asthma symptoms twice a week or more on average in the month prior to study entry
  2. Nocturnal awakening with asthma symptoms more than once per week on average in the month prior to study entry
  3. Two or more emergency department visits, unscheduled physician visits, prednisone courses, or hospitalizations for asthma in the 12 months prior to study entry
  4. Juniper Asthma Control Score (ACS) of 1.25 or greater at the first screening visit
* Absence of GERD symptoms at the time of study entry

Exclusion Criteria:

* Previous anti-reflux or peptic ulcer surgery
* Previous tracheoesophageal fistula repair
* FEV1 less than 60% of predicted normal value at screening visit and as measured immediately before methacholine bronchoprovocation; methacholine bronchoprovocation will be limited to participants with a FEV1 greater than or equal to 70% of predicted value in accordance with American Thoracic Society (ATS) guidelines
* History of a premature birth of less than 33 weeks gestation or any neonate requiring a significant level of respiratory care, including mechanical ventilation
* Any major chronic illness, including but not limited to non-skin cancer, cystic fibrosis, bronchiectasis, myelomeningocele, sickle cell anemia, endocrine disease, congenital heart disease, congestive heart failure, stroke, severe hypertension, insulin-dependent diabetes mellitus, kidney failure, liver disorder, immunodeficiency state, significant neuro-developmental delay or behavioral disorder (excluding mild attention deficit hyperactivity disorder), or other condition that would interfere with participation in the study
* History of phenylketonuria
* Medications for treatment of GI symptoms (e.g., proton pump inhibitors, H2 blockers, bethanechol, metoclopramide) in the month prior to study entry (intermittent anti-acids are allowed)
* Use of theophylline preparations, azoles, anti-coagulants, insulin for Type I diabetes, digitalis, or oral iron supplements when administered for iron deficiency in the month prior to study entry
* Use of any investigative drug in the 2 months prior to study entry
* Previous adverse effects from lansoprazole, other proton pump inhibitors, or sensitivity to aspartame
* Inability or unwillingness of the legal guardian to provide consent
* Inability or unwillingness of the child to provide assent
* Inability to take study medication
* Inability to perform baseline measurements
* Less than 80% completion of screening period diaries
* Inability to contact by telephone
* Planning to move out of the area in the 6 months following study entry
* Pregnancy

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 306 (Actual)
Dates: Start 2007-03; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Holbrook, PhD, MPH, Principal Investigator — Johns Hopkins University School of Public Health; Gerald Teague, MD, Principal Investigator — University of Virginia
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Diego, San Diego, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - University of South Florida College of Medicine, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri, Kansas City School of Medicine, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - North Shore-Long Island Jewish Health System, New Hyde Park, New York
  - New York University School of Medicine, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Davis Heart and Lung Research Institute, Columbus, Ohio
  - Penn Presbyterain Medical Center/Penn Lung Center, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Vermont Lung Center at The University of Vermont, Burlington, Vermont

REFERENCES:
- [Result] Writing Committee for the American Lung Association Asthma Clinical Research Centers; Holbrook JT, Wise RA, Gold BD, Blake K, Brown ED, Castro M, Dozor AJ, Lima JJ, Mastronarde JG, Sockrider MM, Teague WG. Lansoprazole for children with poorly controlled asthma: a randomized controlled trial. JAMA. 2012 Jan 25;307(4):373-81. doi: 10.1001/jama.2011.2035. PMID 22274684
- [Derived] Kaminsky DA, He J, Henderson R, Dixon AE, Irvin CG, Mastronarde J, Smith LJ, Sugar EA, Wise RA, Holbrook JT. Bronchodilator response does not associate with asthma control or symptom burden among patients with poorly controlled asthma. Respir Med. 2023 Nov;218:107375. doi: 10.1016/j.rmed.2023.107375. Epub 2023 Aug 1. PMID 37536444
- [Derived] Lang JE, Holbrook JT, Mougey EB, Wei CY, Wise RA, Teague WG, Lima JJ; American Lung Association-Airways Clinical Research Centers. Lansoprazole Is Associated with Worsening Asthma Control in Children with the CYP2C19 Poor Metabolizer Phenotype. Ann Am Thorac Soc. 2015 Jun;12(6):878-85. doi: 10.1513/AnnalsATS.201408-391OC. PMID 25844821
- [Derived] Fitzpatrick AM, Holbrook JT, Wei CY, Brown MS, Wise RA, Teague WG; American Lung Association's Asthma Clinical Research Centers Network. Exhaled breath condensate pH does not discriminate asymptomatic gastroesophageal reflux or the response to lansoprazole treatment in children with poorly controlled asthma. J Allergy Clin Immunol Pract. 2014 Sep-Oct;2(5):579-86.e7. doi: 10.1016/j.jaip.2014.04.006. Epub 2014 May 21. PMID 25213052
- [Derived] Nguyen JM, Holbrook JT, Wei CY, Gerald LB, Teague WG, Wise RA; American Lung Association Asthma Clinical Research Centers. Validation and psychometric properties of the Asthma Control Questionnaire among children. J Allergy Clin Immunol. 2014 Jan;133(1):91-7.e1-6. doi: 10.1016/j.jaci.2013.06.029. Epub 2013 Aug 6. PMID 23932458
- [Derived] Lima JJ, Lang JE, Mougey EB, Blake KB, Gong Y, Holbrook JT, Wise RA, Teague WG. Association of CYP2C19 polymorphisms and lansoprazole-associated respiratory adverse effects in children. J Pediatr. 2013 Sep;163(3):686-91. doi: 10.1016/j.jpeds.2013.03.017. Epub 2013 Apr 24. PMID 23623526
- [Derived] Mougey E, Lang JE, Allayee H, Teague WG, Dozor AJ, Wise RA, Lima JJ. ALOX5 polymorphism associates with increased leukotriene production and reduced lung function and asthma control in children with poorly controlled asthma. Clin Exp Allergy. 2013 May;43(5):512-20. doi: 10.1111/cea.12076. PMID 23600541
- [Derived] Blake K, Teague WG. Gastroesophageal reflux disease and childhood asthma. Curr Opin Pulm Med. 2013 Jan;19(1):24-9. doi: 10.1097/MCP.0b013e32835b582b. PMID 23197288

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted from April 2007 to April 2011
Groups:
- Lansoprazole Group: 15 mg/day by mouth for children weighing less than 30kg, one tablet per day in the evening before a meal 30 mg/day by mouth for children weighing 30 kg or more, two tablets per day in the evening before a meal
- Placebo Group: Matching placebo with no active ingredients. Either 1 or 2 tablets per day, depending on weight, in the evening before a meal
Period: Overall Study
Arm/Group | Lansoprazole Group | Placebo Group
Started | 157 | 149
Completed | 131 | 132
Not Completed | 26 | 17

BASELINE CHARACTERISTICS:
Groups:
- Lansoprazole Group: 15 mg/day for children weighing less than 30kg 30 mg/day for children weighing 30 kg or more
- Placebo Group: Matching placebo
- Total: Total of all reporting groups
Arm/Group | Lansoprazole Group | Placebo Group | Total
Number analyzed (Participants) | 157 | 149 | 306
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 157 | 149 | 306
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 11 (3) | 11 (3) | 11 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 63 | 118
  Male | 102 | 86 | 188
Region of Enrollment [Number; unit: participants]
  United States | 157 | 149 | 306

OUTCOME MEASURES:

1. Primary Outcome: Change in Juniper Asthma Control Score (ACS)
Description: Score ranges from 0 to 6, a lower score indicated better asthma control. Scores above 1.5 are indicative of poor asthma control; score obtained from questionnaire with 6 questions related to asthma control and FEV (amount of air expired in the first second during a forced expiratory maneuver); number presents an average of the change from baseline to all follow-up points
Time Frame: Measured at Weeks 0, 4, 8, 12, 24
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Lansoprazole Group | Placebo Group
Number analyzed (Participants) | 149 | 157
score | 1.1 [0.9 to 1.2] | 1.0 [0.9 to 1.1]
Statistical Analysis 1: Comparison: Lansoprazole Group vs Placebo Group; All participants included in the analysis. The model includes the data (ACQ scores) from all time points including baseline. The treatment effect (delta-delta) comparing the difference from baseline at 6 months is estimated from the model. Longitudinal models estimated the change from baseline to 6 months in a measurement using generalized estimating equations with an unstructured or exchangeable covariance matrix to adjust for repeated measures; Test type: Superiority or Other; p = 0.12, Regression, Linear; Linear mixed effects model is robust to data that are missing at random that has characteristics similar to multiple imputation techniques; Mean Difference (Net) = 0.2, 95% CI 2-sided [0.0 to 0.3], Standard Error of Mean 0.086

2. Secondary Outcome: Asthma-specific Quality of Life
Description: Scores range from 1 to 7 with higher values indicating better asthma-related quality of life; questionnaire measures functional impairments that are most troublesome to children as a result of their asthma; number presents an average of the change from baseline to all follow-up points
Time Frame: Measured at Weeks 0, 4, 8, 12, 16, 20, 24
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Lansoprazole Group | Placebo Group
Number analyzed (Participants) | 149 | 157
score | 5.8 [5.7 to 6.0] | 6.0 [5.9 to 6.2]
Statistical Analysis 1: Comparison: Lansoprazole Group vs Placebo Group; Test type: Superiority or Other; p = 0.65, Regression, Linear; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.3 to 0.2], Standard Error of Mean 0.2593

3. Secondary Outcome: Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: A measure of pulmonary function, specifically the amount of expired air in the first second during a forced expiratory maneuver while seated; test performed at least 4 hours after last dose of short-acting bronchodilator and at least 12 hours after long-acting bronchodilator; number presents an average of the change from baseline to all follow-up points
Time Frame: Measured at Weeks 0, 4, 8, 12, 16, 20, 24
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Lansoprazole Group | Placebo Group
Number analyzed (Participants) | 149 | 157
Liters | 2.2 [2.1 to 2.4] | 2.3 [2.1 to 2.4]
Statistical Analysis 1: Comparison: Lansoprazole Group vs Placebo Group; Test type: Superiority or Other; p = 0.99, Regression, Linear; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.0906

4. Secondary Outcome: Rate of Episodes of Poor Asthma Control (EPAC)
Description: Episodes of poor asthma control are defined as any one of the following:
  * 2 consecutive days with peak flow at less than 70% of baseline
  * prescription of oral corticosteroids for asthma
  * seeking urgent medical care for asthma symptoms
  EPAC was measured by review of daily diaries that were maintained over the entire course of followup, i.e, 24 weeks
Time Frame: Measured daily for 24 weeks by diary
Population: The number of episodes of poor asthma control that occurred in each group over the 24-week follow-up period. Some participants experienced more than one EPAC over the course of follow-up
Measure: Number; unit: number of episodes of poor asthma contrl
Arm/Group | Lansoprazole Group | Placebo Group
Number analyzed (Participants) | 146 | 149
number of episodes of poor asthma contrl | 230 | 184
Statistical Analysis 1: Comparison: Lansoprazole Group vs Placebo Group; Test type: Superiority or Other; p = 0.30, negative binomial; Risk Ratio (RR) = 1.2, 95% CI 2-sided [0.9 to 1.7]

5. Secondary Outcome: Asthma Symptom Utility Index (ASUI)
Description: ASUI is a utility score that ranges from 0 to 1, with higher values indicating better asthma control; info obtained from questionnaire about asthma symptoms; number presents an average of the change from baseline to all follow-up points
Time Frame: Measured at Weeks 0, 4, 8, 12, 16, 20, 24
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Lansoprazole Group | Placebo Group
Number analyzed (Participants) | 149 | 157
score | 0.86 [0.83 to 0.88] | 0.88 [0.86 to 0.90]
Statistical Analysis 1: Comparison: Lansoprazole Group vs Placebo Group; Test type: Superiority or Other; p = 0.14, Regression, Linear; Model includes the data from all time points. Treatment effect (delta-delta) comparing the difference from baseline at 24 weeks is from the model; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.07 to 0.01], Standard Error of Mean 0.02

6. Secondary Outcome: Airways Reactivity (Assessed by Methacholine PC20)
Description: Presence and degree of airway hyperresponsiveness; change from baseline to 24 weeks for airways reactivity assessed by methacholine post-diluent baseline (PC20) after medication holds
Time Frame: Measured at Weeks 0 and 24
Measure: Mean (95% Confidence Interval); unit: mg/mL
Arm/Group | Lansoprazole Group | Placebo Group
Number analyzed (Participants) | 56 | 63
mg/mL | 2.6 [2.0 to 3.3] | 2.5 [1.7 to 3.4]
Statistical Analysis 1: Comparison: Lansoprazole Group vs Placebo Group; Test type: Superiority or Other; p = 0.20, Regression, Linear; Mean Difference (Net) = -0.8, 95% CI 2-sided [-2.1 to 0.4]

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Adverse event reported at study visits after randomization. Only participants completing at least on follow-up medical history form are included,
Arm/Group | Lansoprazole Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 11/149 | 9/157
Other Adverse Events (participants affected / at risk) | 93/147 | 78/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Lansoprazole Group (N=149) | Placebo Group (N=157)
asthma excerbation (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 5/147 (5)
Vomiting and strep throat (Infections and infestations) | 0 (0) | 1 (1)
Mood disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pneumonia requiring hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Severe constipation (Gastrointestinal disorders) | 0 (0) | 1/1 (1)
Elective surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lansoprazole Group (N=147) | Placebo Group (N=150)
upper respiratory infection (Infections and infestations) | 93 | 74
Sore throat (Respiratory, thoracic and mediastinal disorders) | 77 | 59
Group A streptococcus (Infections and infestations) | 6 | 11
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Otitis media (Ear and labyrinth disorders) | 12 | 10
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 16 | 17

LIMITATIONS AND CAVEATS:
Results limited to patients without overt Gastroesophageal reflux disease(GERD). Did not conduct on-treatment potential hydrogen(pH) probe studies to confirm treatment effect. Protein-pump inhibitors(PPI) dose may not induce maximal acid suppression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No